CLINICAL TRIAL: NCT01265706
Title: 1-year, Prospective, Randomized, Open-label, Parallel Group Observational Study to Evaluate the Safety and Efficacy of 4mg/Day of Pitavastatin Versus 2mg/Day of Pitavastatin in Acute Myocardial Infarction(AMI)
Brief Title: Livalo Acute Myocardial Infarction Study (LAMIS)
Status: Completed | Type: Observational
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: PTV_LAMIS II
Record Dates: First submitted 2010-10-18; First posted 2010-12-23 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Acute Myocardial Infarction
Keywords: Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is performed to observe the incidence of major cardiovascular events in Korean patients with AMI after giving pitavastatin 2mg and 4mg longer than 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI, NSTEMI
* Patients satisfying at least one of the followings

  1. Patients with LDL-C ≥ 130 mg/dL
  2. Patients with LDL-C ≥ 100 mg/dL who are regarded as required cholesterol lowering therapy by the investigator
  3. Patients taking statin are required continuous cholesterol lowering therapy
* Patients satisfying at least two of the followings

  1. The change of Ischemic ECG
  2. CK, CK-MB, Troponin-I increased more than two times
  3. The symptom of ACS

Exclusion Criteria:

1. Patients with in-stent restenosis after PCI or coronary artery bypass
2. Patients with cardiogenic shock
3. Patients with severe heart failure (Left ventricular ejection fraction is less than 30%)
4. Patients who are taking cyclosporine
5. Patients who experienced hypersensitivity to pitavastatin
6. Patients under dialysis treatment
7. Patients who are participating other clinical trials
8. Patients who can not stop taking concomitant drugs
9. Pregnant or lactating women or suspected pregnancy
10. Patients who are regarded as ineligible for this study by the investigator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AMI patients who are in need to be treated by statins
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of TLR-MACE for 1 year after enrollment | 1 year after enrollment

SECONDARY OUTCOMES:
Incidence of TVR-MACE for 1 year after enrollment | 1 year after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Hong, Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea